CLINICAL TRIAL: NCT02097732
Title: Ipilimumab Induction in Patients With Melanoma Brain Metastases Receiving Stereotactic Radiosurgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely due to a change in the standard of care treatment
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2013.114; HUM00082134 (Other: University of Michigan)
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Results first posted 2018-01-19 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Melanoma; Brain Metastases
Keywords: Metastatic melanoma; Brain metastases; Radiation therapy; Immune therapy
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — Ipilimumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B: No induction (Active Comparator): Participants will undergo stereotactic radiosurgery (SRS) followed 2-3 weeks later by ipilimumab, which is given once every 3 weeks for a total of 4 doses.
  Interventions: Drug: Ipilimumab; Procedure: Stereotactic Radiosurgery
- A: Induction (Experimental): Patients will receive 2 doses of ipilimumab, which is given once every 3 weeks, prior to stereotactic radiosurgery (SRS), followed by 2 more doses of ipilimumab, for a total of 4 doses.
  Interventions: Drug: Ipilimumab; Procedure: Stereotactic Radiosurgery

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab 3mg/kg given intravenously over 90 minutes, every 3 weeks for a total of 4 doses.
Procedure: Stereotactic Radiosurgery — Stereotactic radiosurgery is a type of focused radiation therapy. It requires the placement of a metal frame on the head for several hours.

SUMMARY:
This is a study to test the efficacy of using standard immune therapy for melanoma prior to stereotactic radiosurgery (ipilimumab induction), as compared to stereotactic radiosurgery followed by immune therapy. The study's hypothesis is that ipilimumab induction is as good as or better than controlling brain metastases as compared to stereotactic radiosurgery followed by immune therapy.

DETAILED DESCRIPTION:
This is a randomized Phase II selection study investigating the use of ipilimumab induction prior to stereotactic radiosurgery (SRS), versus no induction, for melanoma brain metastases. Participants will be randomized to Arm A "Induction" (two doses of ipilimumab prior to SRS, two doses of ipilimumab after SRS) versus Arm B "No induction" (SRS first, followed by 4 doses of ipilimumab). Participants will undergo multiple dynamic contrast-enhanced MRIs of the brain and submit blood samples for immune testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically-confirmed diagnosis of melanoma who have imaging findings suggestive of 1 to 4 brain metastases
* At least one lesion in the brain that is measurable, which is defined as ≥5 x 5mm (Prior craniotomy and surgical resection is allowed, as long as there is at least one remaining measurable lesion in the brain)
* Patients must be candidates for stereotactic radiosurgery (SRS) and planning to undergo SRS
* Patients must be candidates for ipilimumab as determined by the treating physician
* Patients must be neurologically asymptomatic, or very minimally symptomatic, as judged by the treating physicians
* At least 3 weeks has elapsed from any prior therapy, and the patient has recovered from side effects to ≤ grade 1 toxicities per Common Terminology Criteria (CTC) for Adverse Events
* Age > or = 18 years old
* Performance status of ECOG of 0 or 1 (ECOG is the Eastern Oncology Cooperative Group Scoring system used to quantify cancer patients' general well-being and activities of daily life; scores range from 0 to 5 where 0 is perfect health and 5 is death)
* Adequate organ and marrow function: alanine aminotransferase (ALT ) < 2.5x's upper limit of normal (ULN) of the institutional normal reference range, aspartate aminotransferase (AST) < 2.5x's ULN of the institutional normal reference range, Bilirubin < 1.5x's ULN of the institutional normal reference range, Creatinine < 2.0 milligrams per deciliter, Platelets > 50,000 per microliter
* Women of child-bearing potential must agree to use adequate contraception, defined as complete abstinence from intercourse with men or two methods
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Previous radiotherapy to the lesion(s) of interest, including prior treatment with whole brain radiation therapy (WBRT). Prior treatment with SRS is allowed if the index lesion(s) is in a different, non-contiguous location than the previously treated lesion.
* Patients who have previously received ipilimumab, PD-1 inhibitors or PD-L1 inhibitors are excluded due to the potential of effects on primary outcome
* Patients who require WBRT or surgery at the time of enrollment
* Neurologic symptoms or imaging findings that necessitate the use of steroids on the day of enrollment or in the prior 7 days
* Highly suspicious magnetic resonance imaging (MRI) or cerebrospinal fluid evidence of leptomeningeal metastases, unless all measurable disease is localized and SRS is considered the treatment of choice
* Concurrent treatment with any other anti-neoplastic drug or concurrent participation in another therapeutic clinical trial
* Patients unable to undergo or tolerate MRI scans (presence of cardiac pacemaker, implanted cardiac defibrillator, aneurysm clips, history of allergic reaction/hypersensitivity to gadolinium)
* Women who are pregnant or are nursing
* Patients with absolute lymphocyte count of <500 cells/microliter, who are known to be HIV positive, who have clinically significant active autoimmune disease, or are receiving immunosuppression following solid organ or stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lao, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | B: No Induction | A: Induction
Started | 1 | 3
Completed | 1 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B: No Induction | A: Induction | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Continuous [Mean (Full Range); unit: years] | 69 [69 to 69] | 55 [48 to 62] | 58 [48 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Local Control Rate
Description: The number of patients in each arm who are free from progression in the index (radiated) lesions in the brain at 6 months.
  Immune related response criteria was used to assess response to treatment. Immune-related Progressive Disease (irPD) in this trial is defined as an increase in tumor burden ≥25% relative to nadir (minimum recorded tumor burden), with confirmation by a repeat, consecutive assessment no less than 4 weeks from the date first documented.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | B: No Induction | A: Induction
Number analyzed (Participants) | 1 | 3
Participants | 1 | 3

2. Secondary Outcome: Overall Survival Rate
Description: Number of participants alive at 5 years after enrollment.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Groups:
- B: No Induction: Participants will undergo stereotactic radiosurgery (SRS) followed 2-3 weeks later by ipilimumab, which is given once every 3 weeks for a total of 4 doses. Ipilimumab: Ipilimumab 3mg/kg given intravenously over 90 minutes, every 3 weeks for a total of 4 doses. Stereotactic Radiosurgery: Stereotactic radiosurgery is a type of focused radiation therapy. It requires the placement of a metal frame on the head for several hours.
- A: Induction: Patients will receive 2 doses of ipilimumab, which is given once every 3 weeks, prior to stereotactic radiosurgery (SRS), followed by 2 more doses of ipilimumab, for a total of 4 doses. Ipilimumab: Ipilimumab 3mg/kg given intravenously over 90 minutes, every 3 weeks for a total of 4 doses. Stereotactic Radiosurgery: Stereotactic radiosurgery is a type of focused radiation therapy. It requires the placement of a metal frame on the head for several hours.
Arm/Group | B: No Induction | A: Induction
Number analyzed (Participants) | 1 | 3
participants | 1 | 2

3. Secondary Outcome: Regional (Intracranial) Control Rate
Description: The proportion of patients in each arm who are free from progression in the index (radiated) lesions and free from new brain metastases at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | B: No Induction | A: Induction
Number analyzed (Participants) | 1 | 3
Participants | 1 | 3

4. Secondary Outcome: Intracranial Response Rate
Description: Response of treated (irradiated) brain metastases to combination therapy with ipilimumab and stereotactic radiosurgery using immune-related response criteria.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | B: No Induction | A: Induction
Number analyzed (Participants) | 1 | 3
Participants | 1 | 3

5. Secondary Outcome: Time to Progression
Description: Time to progression in the brain due to treated metastases or new brain metastases. Immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) was used to assess response. Progression was defined as an increase in tumor burden ≥25% relative to nadir (minimum recorded tumor burden), with confirmation by a repeat, consecutive assessment no less than 4 wk from the date first documented.
Time Frame: From date of enrollment to up to 2 years
Population: Of the 4 patients, 2 patients remained progression-free throughout the 2-year time frame for data collection for this outcome measure.
Measure: Number; unit: participants
Arm/Group | B: No Induction | A: Induction
Number analyzed (Participants) | 1 | 3
participants
  5 months, 27 days | 0 | 1
  19 months, 3 days | 1 | 0

6. Other Pre Specified Outcome: Imaging Correlates on Dynamic-contrast Enhanced MRI of the Brain
Description: Exploratory endpoints: Interval changes in dynamic MRI parameters such as perfusion, blood volume, vascular permeability (Ktrans), and diffusion tensor imaging; the change in 3D tumor volume.
Time Frame: 6 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Immune Correlates
Description: Exploratory endpoints: Interval changes in immune markers in the blood
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 6 months after study start. All-cause mortality is observed up to 5 years.
Description: Both arms were combined in the reporting of Adverse Events because both arms received the same two interventions.
Groups:
- Ipilimumab and SRS: (Induction) Patients will receive 2 doses of ipilimumab, which is given once every 3 weeks, prior to stereotactic radiosurgery (SRS), followed by 2 more doses of ipilimumab, for a total of 4 doses.
  OR
  (No Induction) Participants will undergo stereotactic radiosurgery (SRS) followed 2-3 weeks later by ipilimumab, which is given once every 3 weeks for a total of 4 doses.
  Ipilimumab: Ipilimumab 3mg/kg given intravenously over 90 minutes, every 3 weeks for a total of 4 doses.
  Stereotactic Radiosurgery: Stereotactic radiosurgery is a type of focused radiation therapy. It requires the placement of a metal frame on the head for several hours.
Arm/Group | Ipilimumab and SRS
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab and SRS (N=4)
Alanine aminotransferase increased (Investigations) | 1 (1)
Concentration impairment (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Edema limbs (Vascular disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Flu like symptoms (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hot flashes (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Decreased T4 (Investigations) | 1 (1)
Vitamin D Deficiency (Investigations) | 1 (1)
Low Testosterone (Investigations) | 1 (2)
Elevated LDH (Investigations) | 1 (2)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (2)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Periorbital edema (Vascular disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study halted prematurely due to a change in the standard of care treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes